CLINICAL TRIAL: NCT05766852
Title: Potential Benefits of the Somatic Psychoeducational Intervention for Improving the Health and Wellness of Healthcare Providers
Brief Title: Potential Benefits of the Somatic Psychoeducational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202200233
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-06

CONDITIONS: Work Related Stress
Keywords: Polyvagal Theory; Stress; Trauma; Neuroendocrine biomarkers; Somatic interventions; Oxytocin; Vasopressin; PTSD; Mental health; Neuroendocrine functioning; professional health; Physical health; Emotional health; Coping behaviors; Mindfulness; Burnout; Tai Chi; Psychoeducation; Breathing exercises; healthcare providers
MeSH Terms: conditions — Occupational Stress; Wounds and Injuries; Diabetes Insipidus; Stress Disorders, Post-Traumatic; Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to Group A or Group B and either Monday or Thursday class according to their availability. Participants who are not able to attend either Monday or Thursday will have the option to complete the intervention virtually. Intervention Group A will be provided the intervention including breath and psychoeducation and Group B will be provided the intervention including breath, movement, and psychoeducation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Breath + Psychoeducation (Active Comparator): Participants will be asked to participate in the 3 1.5-hour intervention classes. The pre-intervention and post-intervention assessments will require participants to complete a 20-25-minute online survey via Qualtrics and provide saliva samples.
  Interventions: Behavioral: Somatic Psychoeducational Intervention
- Group B: Breath + Movement + Psychoeducation (Experimental): Participants will be asked to participate in the 3 1.5-hour intervention classes. The pre-intervention and post-intervention assessments will require participants to complete a 20-25-minute online survey via Qualtrics and provide saliva samples.
  Interventions: Behavioral: Somatic Psychoeducational Intervention

INTERVENTIONS:
Behavioral: Somatic Psychoeducational Intervention — Participants will work on increasing bodily awareness by learning psychoeducation, movement techniques, and relaxation.

SUMMARY:
The goal of this clinical trial is to explore possible benefits and mechanisms through which the Somatic Psychoeducational Intervention can improve health and wellness in health care providers (HCP). The main goals of the study are:

* To understand how the participants are doing with regard to their mindfulness, coping behaviors, emotional, physical, and work health, and autonomic reactivity (the degree participants physiologically respond).
* To investigate whether pre-intervention measures relate to the overall functioning of the HCPs.
* To determine the 1-week and 1-month post-intervention effects of the Intervention(s)
* To identify individual characteristics that influence the effectiveness of the intervention at the 1-week and 1-month post-intervention assessments.

Participants will:

* complete the online pre-assessment measures regarding how they are doing emotionally and with respect to their work situation.
* complete pre-intervention, 1-week post-intervention, and 1-month post-intervention assessments that involve completion of online measures and collection of saliva samples.
* participated in the intervention (which involves 4.5 hours; the 1.5-hour classes will be administered over three weeks).

Researchers will compare the Intervention Group A to Intervention Groub B to see if the Intervention Group B experiences greater improvements in their health and wellness.

DETAILED DESCRIPTION:
It is the intent of this proposal to experimentally explore in health care providers (HCP) the possible benefits and mechanisms through which the Somatic Psychoeducational Intervention can influence emotional and physical health and autonomic and neuroendocrine functioning. This will be accomplished by our team by using well-validated self-report measures of mental health and autonomic reactivity and non-invasive measurements of levels of oxytocin.

Specific Aims:

* Specific Aim 1: To understand via the screening online assessment how the participants are doing with regard to their mindfulness, coping behaviors, emotional, physical, and work health, and self-reported autonomic reactivity
* Specific Aim 2: To investigate whether pre-intervention measures of autonomic reactivity and the neuropeptides oxytocin relate to the overall functioning of the HCPs.
* Specific Aim 3: To determine if the intervention leads to improvements in functioning 1-week and 1-month post the Intervention
* Specific Aim 4: To identify individual characteristics that influence the effectiveness of the intervention 1-week and 1-month post intervention.

Experimental design

* In the Screening Phase, we will recruit healthcare providers, starting with bedside nurses. We will make available a link to the study so that participants could complete the online pre-assessment measures regarding how they are doing emotionally and with respect to their work situation.
* In the Intervention Phase, the participants will be assigned to either Group A or Group B based on their provided availability. Participants who are unable to attend the in-person intervention will be invited to complete the pre-recorded intervention virtually. Intervention Group A, which will be provided the intervention including breath and psychoeducation, and Group B, which will be provided the intervention including breath, movement, and psychoeducation.
* The invited participants will complete assessments 1 week before starting the assessment and 1 week after the intervention that involve online measure and collection of saliva samples.
* The Somatic Psychoeducational Intervention will be provided in three 1.5-hour classes and the participants will be awarded for their participation financially and through continuing education credits.
* In addition, the participants will complete the online 1-month post-intervention assessment
* Between-subject analyses will compare the session 1 data to determine if the participants in Group B exhibit greater improvements than the participants in Intervention Group A. Within-subject repeated measures analyses will determine the potential benefits of the intervention for all participants by comparing their functioning at the various time points.

  * For the outcome measures, change scores will be calculated to determine the change from the pre-intervention to the 1-week post-intervention assessment, and from the 1-week post-intervention assessment to the 1-month post-intervention assessment. These changes scores will be used to determine if there are pre-intervention factors that impact the success of the intervention.

ELIGIBILITY:
Inclusion Criteria:

-Individuals are eligible to participate in Screening Phase of the study if they are at least 18 years old and are bedside nurses in units at the 8th street location or North Campus of the University of Florida Health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Measuring Change in Depressive Symptoms using the Patient Health Questionnaire (PHQ-8) self-report questionnaire. | Baseline up to 1-month (post-intervention)
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) will be used to assess current depression. Depression can be defined as ongoing feelings of sadness or loss of interest in typically pleasurable activities. This measure includes 8 items that are answered via a 4-point Likert scales (0 = not at all, 1 = several days, 2 = more than half the days, and 3 - nearly every day). Total scores range from 0 to 24, with higher indicated more symptoms of depression.
Change in autonomic reactivity using the Body Perception Questionnaire self-report questionnaire. | Baseline up to 1-month (post-intervention)
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Measuring Change in anxiety using the General Anxiety Disorder 7 self-report questionnaire. | Baseline up to 1-month (post-intervention)
  This 7-item measure is scored on a 4-point Likert scale (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Items are summed, with the higher scores indicating increased symptoms of anxiety.
Measuring Change in social engagement using the Neuroception of Psychological Safety Scale self-report questionnaire. | Baseline up to 1-month (post-intervention)
  This 14-item measure is scored on a 5-point Likert scale (Strongly Disagree = 1 to Strongly Agree = 5). Items are summed, with the higher scores indicating greater social engagement.
Measuring Change in Posttraumatic Stress Symptoms using the Posttraumatic Stress Disorder Checklist 5 self-report questionnaire. | Baseline up to 1-month (post-intervention)
  This 8-item measure scored on a 5-point Likert scale (not at all = 0 to extremely = 4). Items are summed, with the higher scores indicating increased symptoms are depression.
Measuring Change in Mindfulness using the Five Facets of Mindfulness self-report questionnaire. | Baseline up to 1-month (post-intervention)
  This 15-item measure assess mindfulness via a 5-point Likert scale (Never or very rarely true = 1 to Very often or always true = 5). Higher sum scores are representative of greater mindfulness.
Measuring impact of prior adversity using the Adverse and Traumatic Experiences Scale self-report questionnaire. | Baseline
  This 30-item measure asks about prior adversity (i.e., Childhood adversity, caregiver maltreatment, non-caregiver maltreatment, life-threatening situations, and sudden losses). Participants indicate how impacted they were via a 5-point Likert scale (0 = event did not occur, 1 = occurred and no impact on my life, 2 = minimal impact on my life, 3 = some impact on my life, and 4 = big impact on my life). Higher sum scores are indicative of greater prior adversity.
Measuring change of professional health outcomes using self-report questionnaires. | Baseline up to 1-month (post-intervention)
  Professional fulfillment and Burnout was assessed via the 16-item Professional Fulfillment Index (Professional Fulfillment 6 items, Burnout [Work Exhaustion 4 items and Interpersonal Disengagement 6 items]). Participants indicate how true 6 items assessing Professional Fulfillment are via a 5-point Likert scale (0 = not at all true to 4 = completely true). Higher sum scores are indicative of greater Professional Fulfillment. Participants indicate the degree they have experienced 10 items assessing burnout are via a 5-point Likert scale (0 = not at all to 4 = extremely). Higher sum scores are indicative of increased burnout.
Measuring change in physical stress | Baseline up to 1-month (post-intervention)
  This 9-item measure is scored via a 5-point Likert scale (0 = never to 4 = always). Higher sum scores represent increased physical stress
Measuring change in salivary oxytocin levels via Enzyme Immunoassay kit | Baseline up to 1-month (post-intervention)
  Saliva samples were collected via a passive drool method using Thermo Scientific™ SpeciMAX™ Saliva Collection Tube (Catalog number A50696). Salivary oxytocin concentrates (pg/mL) determined via Enzyme Immunoassay kit (ELISA; Arbor Assays Catalog #K048-H1).

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P Dale, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alleyne S, Dale L, Robertson-Blackmore E, Kishore A, Cuffe S, Fallucco E. United States of America Child and Adolescent Psychiatrists' Career Satisfaction by Career Stage. Acad Psychiatry. 2022 Aug;46(4):441-450. doi: 10.1007/s40596-021-01577-x. Epub 2022 Jan 16. PMID 35034337
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Barello S, Palamenghi L, Graffigna G. Burnout and somatic symptoms among frontline healthcare professionals at the peak of the Italian COVID-19 pandemic. Psychiatry Res. 2020 Aug;290:113129. doi: 10.1016/j.psychres.2020.113129. Epub 2020 May 27. PMID 32485487
- [Background] Baribeau DA, Anagnostou E. Oxytocin and vasopressin: linking pituitary neuropeptides and their receptors to social neurocircuits. Front Neurosci. 2015 Sep 24;9:335. doi: 10.3389/fnins.2015.00335. eCollection 2015. PMID 26441508
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya yogic breathing in the treatment of stress, anxiety, and depression: part I-neurophysiologic model. J Altern Complement Med. 2005 Feb;11(1):189-201. doi: 10.1089/acm.2005.11.189. PMID 15750381
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya Yogic breathing in the treatment of stress, anxiety, and depression. Part II--clinical applications and guidelines. J Altern Complement Med. 2005 Aug;11(4):711-7. doi: 10.1089/acm.2005.11.711. PMID 16131297
- [Background] Cabrera A, Kolacz J, Pailhez G, Bulbena-Cabre A, Bulbena A, Porges SW. Assessing body awareness and autonomic reactivity: Factor structure and psychometric properties of the Body Perception Questionnaire-Short Form (BPQ-SF). Int J Methods Psychiatr Res. 2018 Jun;27(2):e1596. doi: 10.1002/mpr.1596. Epub 2017 Nov 28. PMID 29193423
- [Background] Carter CS, Kenkel WM, MacLean EL, Wilson SR, Perkeybile AM, Yee JR, Ferris CF, Nazarloo HP, Porges SW, Davis JM, Connelly JJ, Kingsbury MA. Is Oxytocin "Nature's Medicine"? Pharmacol Rev. 2020 Oct;72(4):829-861. doi: 10.1124/pr.120.019398. PMID 32912963
- [Background] Carter CS, Grippo AJ, Pournajafi-Nazarloo H, Ruscio MG, Porges SW. Oxytocin, vasopressin and sociality. Prog Brain Res. 2008;170:331-6. doi: 10.1016/S0079-6123(08)00427-5. PMID 18655893
- [Background] Carter CS. Oxytocin pathways and the evolution of human behavior. Annu Rev Psychol. 2014;65:17-39. doi: 10.1146/annurev-psych-010213-115110. Epub 2013 Sep 19. PMID 24050183
- [Background] Carter CS, Pournajafi-Nazarloo H, Kramer KM, Ziegler TE, White-Traut R, Bello D, Schwertz D. Oxytocin: behavioral associations and potential as a salivary biomarker. Ann N Y Acad Sci. 2007 Mar;1098:312-22. doi: 10.1196/annals.1384.006. PMID 17435137
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Cash M, Whittingham K. What facets of mindfulness contribute to psychological well-being and depressive, anxious, and stress-related symptomatology? Mindfulness. 2010;1(3):177-182.
- [Background] Champely, S. (2020). Basic Functions for Power Analysis. R package version 1.3-0, https://CRAN.R-project.org/package=pwr.
- [Background] Cochran DM, Fallon D, Hill M, Frazier JA. The role of oxytocin in psychiatric disorders: a review of biological and therapeutic research findings. Harv Rev Psychiatry. 2013 Sep-Oct;21(5):219-47. doi: 10.1097/HRP.0b013e3182a75b7d. PMID 24651556
- [Background] Coffey KA, Hartman M. Mechanisms of action in the inverse relationship between mindfulness and psychological distress. Complement Health Pract Rev. 2008;13(2):79-91.
- [Background] Dale LP, Bossemeyer Biernacki N, Nunez LV, Herman MS, Turpeau MC, Lange LJ. Factors affecting emotional distress in college students during COVID-19. Manuscript under review by the Journal of American College Health. 2022.
- [Background] Dale LP, Carroll LE, Galen G, Hayes JA, Webb KW, Porges SW. Abuse history is related to autonomic regulation to mild exercise and psychological wellbeing. Appl Psychophysiol Biofeedback. 2009 Dec;34(4):299-308. doi: 10.1007/s10484-009-9111-4. Epub 2009 Aug 26. PMID 19707870
- [Background] Dale LP, Cuffe SP, Sambuco N, Guastello AD, Leon KG, Nunez LV, Bhullar A, Allen BR, Mathews CA. Morally Distressing Experiences, Moral Injury, and Burnout in Florida Healthcare Providers during the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Nov 24;18(23):12319. doi: 10.3390/ijerph182312319. PMID 34886045
- [Background] Dale LP, Cuffe SP, Kolacz J, Leon KG, Bossemeyer Biernacki N, Bhullar A, Nix EJ, Porges SW. Increased Autonomic Reactivity and Mental Health Difficulties in COVID-19 Survivors: Implications for Medical Providers. Front Psychiatry. 2022 May 25;13:830926. doi: 10.3389/fpsyt.2022.830926. eCollection 2022. PMID 35693957
- [Background] Dale LP, Davidson C, Kolacz J. (2020). The Adverse and Traumatic Experiences Scale.
- [Background] Dale LP, Fasciano LC, Shaikh SK, Little Hodge AL, Gracia B, Majdick JM, et al. Maltreatment History and Physiological Regulation in Response to Physical and Emotional Stressors. In S. W. Porges, L. P. Dale, & J. Kolacz. Trauma through the lens of the Polyvagal Theory: Implications for understanding mechanisms and optimizing outcomes. Workshop presentation at 25th Annual International Trauma Conference, Boston, MA.
- [Background] Dale LP, Shaikh SK, Fasciano LC, Watorek VD, Heilman KJ, Porges SW. College females with maltreatment histories have atypical autonomic regulation and poor psychological wellbeing. Psychol Trauma. 2018 Jul;10(4):427-434. doi: 10.1037/tra0000342. Epub 2017 Nov 20. PMID 29154592
- [Background] Doussard-Roosevelt JA, Porges SW. The role of neurobehavioral organization in stress responses: A polyvagal model. 1999.
- [Background] Ellis BJ, Horn AJ, Carter CS, van IJzendoorn MH, Bakermans-Kranenburg MJ. Developmental programming of oxytocin through variation in early-life stress: Four meta-analyses and a theoretical reinterpretation. Clin Psychol Rev. 2021 Jun;86:101985. doi: 10.1016/j.cpr.2021.101985. Epub 2021 Feb 15. PMID 33770582
- [Background] Figueroa MA, Demeersman RE, Manning J. The autonomic and rate pressure product responses of tai chi practitioners. N Am J Med Sci. 2012 Jun;4(6):270-5. doi: 10.4103/1947-2714.97208. PMID 22754878
- [Background] Friedman MJ. Acknowledging the psychiatric cost of war. N Engl J Med. 2004 Jul 1;351(1):75-7. doi: 10.1056/NEJMe048129. No abstract available. PMID 15229311
- [Background] Goelz DV. Tai chi and its effect on post-traumatic stress. Doctoral thesis. The Chicago School of Professional Psychology; 2015
- [Background] Grahn P, Ottosson J, Uvnas-Moberg K. The Oxytocinergic System as a Mediator of Anti-stress and Instorative Effects Induced by Nature: The Calm and Connection Theory. Front Psychol. 2021 Jul 5;12:617814. doi: 10.3389/fpsyg.2021.617814. eCollection 2021. PMID 34290636
- [Background] Grodin MA, Piwowarczyk L, Fulker D, Bazazi AR, Saper RB. Treating survivors of torture and refugee trauma: a preliminary case series using qigong and t'ai chi. J Altern Complement Med. 2008 Sep;14(7):801-6. doi: 10.1089/acm.2007.0736. PMID 18803491
- [Background] Groenewegen PP, Gress S, Schafer W. General Practitioners' Participation in a Large, Multicountry Combined General Practitioner-Patient Survey: Recruitment Procedures and Participation Rate. Int J Family Med. 2016;2016:4929432. doi: 10.1155/2016/4929432. Epub 2016 Mar 7. PMID 27047689
- [Background] Groth SW. Honorarium or coercion: use of incentives for participants in clinical research. J N Y State Nurses Assoc. 2010 Spring-Summer;41(1):11-3; quiz 22. PMID 20882821
- [Background] Guastello AD, Brunson JC, Sambuco N, Dale LP, Tracy NA, Allen BR, Mathews CA. Predictors of professional burnout and fulfilment in a longitudinal analysis on nurses and healthcare workers in the COVID-19 pandemic. J Clin Nurs. 2024 Jan;33(1):288-303. doi: 10.1111/jocn.16463. Epub 2022 Aug 10. PMID 35949164
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Asch DA. Empirical assessment of whether moderate payments are undue or unjust inducements for participation in clinical trials. Arch Intern Med. 2004 Apr 12;164(7):801-3. doi: 10.1001/archinte.164.7.801. PMID 15078651
- [Background] Holst Y, Thorell LB. Adult executive functioning inventory (ADEXI): Validity, reliability, and relations to ADHD. Int J Methods Psychiatr Res. 2018 Mar;27(1):e1567. doi: 10.1002/mpr.1567. Epub 2017 May 12. PMID 28497641
- [Background] Holst Y, Thorell LB. Neuropsychological Functioning in Adults With ADHD and Adults With Other Psychiatric Disorders. J Atten Disord. 2017 Jan;21(2):137-148. doi: 10.1177/1087054713506264. Epub 2016 Jul 28. PMID 24134875
- [Background] Hruska B, Barduhn MS. Dynamic psychosocial risk and protective factors associated with mental health in Emergency Medical Service (EMS) personnel. J Affect Disord. 2021 Mar 1;282:9-17. doi: 10.1016/j.jad.2020.12.130. Epub 2020 Dec 28. PMID 33387746
- [Background] Jones JL, Ackerman D, Barona J, Calle M, Andersen CJ, Kim JE, Volek JS, McIntosh M, Najm W, Lerman RH, Fernandez ML. A Mediterranean low-glycemic-load diet alone or in combination with a medical food improves insulin sensitivity and reduces inflammation in women with metabolic syndrome. British Journal of Medicine & Medical Research. 2011;1(4).
- [Background] Jones JL, Comperatore M, Barona J, Calle MC, Andersen C, McIntosh M, Najm W, Lerman RH, Fernandez ML. A Mediterranean-style, low-glycemic-load diet decreases atherogenic lipoproteins and reduces lipoprotein (a) and oxidized low-density lipoprotein in women with metabolic syndrome. Metabolism. 2012 Mar;61(3):366-72. doi: 10.1016/j.metabol.2011.07.013. Epub 2011 Sep 23. PMID 21944261
- [Background] Joyce S, Shand F, Lal TJ, Mott B, Bryant RA, Harvey SB. Resilience@Work Mindfulness Program: Results From a Cluster Randomized Controlled Trial With First Responders. J Med Internet Res. 2019 Feb 19;21(2):e12894. doi: 10.2196/12894. PMID 30777846
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Khalsa SS, Lapidus RC. Can Interoception Improve the Pragmatic Search for Biomarkers in Psychiatry? Front Psychiatry. 2016 Jul 25;7:121. doi: 10.3389/fpsyt.2016.00121. eCollection 2016. PMID 27504098
- [Background] Keck ME. Corticotropin-releasing factor, vasopressin and receptor systems in depression and anxiety. Amino Acids. 2006 Oct;31(3):241-50. doi: 10.1007/s00726-006-0333-y. Epub 2006 May 29. PMID 16733617
- [Background] Kumsta R, Heinrichs M. Oxytocin, stress and social behavior: neurogenetics of the human oxytocin system. Curr Opin Neurobiol. 2013 Feb;23(1):11-6. doi: 10.1016/j.conb.2012.09.004. Epub 2012 Oct 4. PMID 23040540
- [Background] Kolacz J, Dale LP, Nix EJ, Roath OK, Lewis GF, Porges SW. Adversity History Predicts Self-Reported Autonomic Reactivity and Mental Health in US Residents During the COVID-19 Pandemic. Front Psychiatry. 2020 Oct 27;11:577728. doi: 10.3389/fpsyt.2020.577728. eCollection 2020. PMID 33192715
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lahn MJ. Indices of heart rate variability and compassion in healthcare professionals following stress resilience training [ProQuest Information & Learning]. In Dissertation Abstracts International: Section B: The Sciences and Engineering (Vol. 75, Issue 11-B(E)). 2015
- [Background] Lan C. Tai chi improves natural harmony in autonomic function. N Am J Med Sci. 2012 Jun;4(6):276-7. No abstract available. PMID 22754879
- [Background] Lawn S, Roberts L, Willis E, Couzner L, Mohammadi L, Goble E. The effects of emergency medical service work on the psychological, physical, and social well-being of ambulance personnel: a systematic review of qualitative research. BMC Psychiatry. 2020 Jul 3;20(1):348. doi: 10.1186/s12888-020-02752-4. PMID 32620092
- [Background] Leavitt, K.S. Pat Ogden, Kekuni Minton and Clare Pain, Trauma and the body: A sensorimotor approach to psychotherapy. Clin Soc Work J. 2008;36:221-223.
- [Background] Lewis GF, Hourani L, Tueller S, Kizakevich P, Bryant S, Weimer B, Strange L. Relaxation training assisted by heart rate variability biofeedback: Implication for a military predeployment stress inoculation protocol. Psychophysiology. 2015 Sep;52(9):1167-74. doi: 10.1111/psyp.12455. Epub 2015 Jun 11. PMID 26095854
- [Background] McDonald MA, Yang Y, Lancaster CL. The association of distress tolerance and mindful awareness with mental health in first responders. Psychol Serv. 2022;19(Suppl 1):34-44. doi: 10.1037/ser0000588. Epub 2021 Oct 28. PMID 34726457
- [Background] Meyer-Lindenberg A, Domes G, Kirsch P, Heinrichs M. Oxytocin and vasopressin in the human brain: social neuropeptides for translational medicine. Nat Rev Neurosci. 2011 Aug 19;12(9):524-38. doi: 10.1038/nrn3044. PMID 21852800
- [Background] Minassian A, Maihofer AX, Baker DG, Nievergelt CM, Geyer MA, Risbrough VB; Marine Resiliency Study Team. Association of Predeployment Heart Rate Variability With Risk of Postdeployment Posttraumatic Stress Disorder in Active-Duty Marines. JAMA Psychiatry. 2015 Oct;72(10):979-86. doi: 10.1001/jamapsychiatry.2015.0922. PMID 26353072
- [Background] Morton L, Cogan N, Kolacz J, Calderwood C, Nikolič M, Bacon T, et al. Developing a standardised measure of psychological safety. 35th Annual Conference of the European Health Psychology Society.2021
- [Background] Mosheva M, Gross R, Hertz-Palmor N, Hasson-Ohayon I, Kaplan R, Cleper R, Kreiss Y, Gothelf D, Pessach IM. The association between witnessing patient death and mental health outcomes in frontline COVID-19 healthcare workers. Depress Anxiety. 2021 Apr;38(4):468-479. doi: 10.1002/da.23140. Epub 2021 Feb 5. PMID 33544405
- [Background] Nash WP, Marino Carper TL, Mills MA, Au T, Goldsmith A, Litz BT. Psychometric evaluation of the Moral Injury Events Scale. Mil Med. 2013 Jun;178(6):646-52. doi: 10.7205/MILMED-D-13-00017. PMID 23756071
- [Background] Neumann ID, Landgraf R. Balance of brain oxytocin and vasopressin: implications for anxiety, depression, and social behaviors. Trends Neurosci. 2012 Nov;35(11):649-59. doi: 10.1016/j.tins.2012.08.004. Epub 2012 Sep 11. PMID 22974560
- [Background] Norman SB, Feingold JH, Kaye-Kauderer H, Kaplan CA, Hurtado A, Kachadourian L, Feder A, Murrough JW, Charney D, Southwick SM, Ripp J, Peccoralo L, Pietrzak RH. Moral distress in frontline healthcare workers in the initial epicenter of the COVID-19 pandemic in the United States: Relationship to PTSD symptoms, burnout, and psychosocial functioning. Depress Anxiety. 2021 Oct;38(10):1007-1017. doi: 10.1002/da.23205. Epub 2021 Jul 22. PMID 34293236
- [Background] Papazoglou K. The examination of different pathways leading towards police traumatization: Exploring the role of moral injury and personality in police compassion fatigue [ProQuest Information & Learning]. In Dissertation Abstracts International: Section B: The Sciences and Engineering (Vol. 79, Issue 3-B(E)). 2018
- [Background] Perez LG, Abrams MP, Lopez-Martinez AE, Asmundson GJ. Trauma exposure and health: the role of depressive and hyperarousal symptoms. J Trauma Stress. 2012 Dec;25(6):641-8. doi: 10.1002/jts.21762. Epub 2012 Nov 26. PMID 23184401
- [Background] Phillips KFV, Power MJ. A new self-report measure of emotion regulation in adolescents: The Regulation of Emotions Questionnaire, Clin Psychol Psychother. 2007;14(2):145-156.
- [Background] Porges SW. Neuroception: A subconscious system for detecting threats and safety. Zero Three. 2004; 24(5):19-24.
- [Background] Porges, SW. Polyvagal Safety: Attachment, Communication, Self-Regulation. WW Norton & Company; 2021.
- [Background] Porges SW. Stress and parasympathetic control. Stress science: neuroendocrinology. 2010 Apr 6:306-12.2010
- [Background] Porges SW. Body Perception Questionnaire Short Form© 1993, 2015
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Porges SW. The polyvagal theory: neurophysiological foundations of emotions, attachment, communication, and self-regulation (Norton Series on Interpersonal Neurobiology). WW Norton & Company; 2011 Apr 25.
- [Background] Porges SW. The Polyvagal Theory: phylogenetic contributions to social behavior. Physiol Behav. 2003 Aug;79(3):503-13. doi: 10.1016/s0031-9384(03)00156-2. PMID 12954445
- [Background] Porges SW. The polyvagal theory: phylogenetic substrates of a social nervous system. Int J Psychophysiol. 2001 Oct;42(2):123-46. doi: 10.1016/s0167-8760(01)00162-3. PMID 11587772
- [Background] Price CJ, Hooven C. Interoceptive Awareness Skills for Emotion Regulation: Theory and Approach of Mindful Awareness in Body-Oriented Therapy (MABT). Front Psychol. 2018 May 28;9:798. doi: 10.3389/fpsyg.2018.00798. eCollection 2018. PMID 29892247
- [Background] Price M, Szafranski DD, van Stolk-Cooke K, Gros DF. Investigation of abbreviated 4 and 8 item versions of the PTSD Checklist 5. Psychiatry Res. 2016 May 30;239:124-30. doi: 10.1016/j.psychres.2016.03.014. Epub 2016 Mar 8. PMID 27137973
- [Background] Romano A, Tempesta B, Micioni Di Bonaventura MV, Gaetani S. From Autism to Eating Disorders and More: The Role of Oxytocin in Neuropsychiatric Disorders. Front Neurosci. 2016 Jan 12;9:497. doi: 10.3389/fnins.2015.00497. eCollection 2015. PMID 26793046
- [Background] Russell ML, Moralejo DG, Burgess ED. Paying research subjects: participants' perspectives. J Med Ethics. 2000 Apr;26(2):126-30. doi: 10.1136/jme.26.2.126. PMID 10786324
- [Background] Sayer NA, Spoont M, Murdoch M, Parker LE, Hintz S, Rosenheck R. A qualitative study of U.S. veterans' reasons for seeking Department of Veterans Affairs disability benefits for posttraumatic stress disorder. J Trauma Stress. 2011 Dec;24(6):699-707. doi: 10.1002/jts.20693. Epub 2011 Nov 22. PMID 22109077
- [Background] Schmid RF, Thomas J. The interactive effects of heart rate variability and mindfulness on indicators of well-being in healthcare professionals' daily working life. Int J Psychophysiol. 2021 Jun;164:130-138. doi: 10.1016/j.ijpsycho.2021.01.012. Epub 2021 Feb 3. PMID 33548348
- [Background] Schoniger C, Braun D, Siepmann M, Petrowski K. Comparison of the HRV of Emergency Physicians in the HEMS During Helicopter Operations: Analysis of Differences as a Function of Number of Operations and Workload. Appl Psychophysiol Biofeedback. 2020 Dec;45(4):249-257. doi: 10.1007/s10484-020-09480-1. PMID 32627104
- [Background] Schulz-Heik RJ, Meyer H, Mahoney L, Stanton MV, Cho RH, Moore-Downing DP, Avery TJ, Lazzeroni LC, Varni JM, Collery LM, Bayley PJ. Results from a clinical yoga program for veterans: yoga via telehealth provides comparable satisfaction and health improvements to in-person yoga. BMC Complement Altern Med. 2017 Apr 4;17(1):198. doi: 10.1186/s12906-017-1705-4. PMID 28376861
- [Background] Shin HJ, Rosen CS, Greenbaum MA, Jain S. Longitudinal correlates of aggressive behavior in help-seeking U.S. veterans with PTSD. J Trauma Stress. 2012 Dec;25(6):649-56. doi: 10.1002/jts.21761. PMID 23225031
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Slattery DA, Neumann ID. Oxytocin and Major Depressive Disorder: Experimental and Clinical Evidence for Links to Aetiology and Possible Treatment. Pharmaceuticals (Basel). 2010 Mar 16;3(3):702-724. doi: 10.3390/ph3030702. PMID 27713275
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Background] van der Kolk BA. Clinical implications of neuroscience research in PTSD. Ann N Y Acad Sci. 2006 Jul;1071:277-93. doi: 10.1196/annals.1364.022. PMID 16891578
- [Background] Van der Kolk, B. Posttraumatic therapy in the age of neuroscience. Psychoanalytic dialogues. 2002;12(3): 381-392.
- [Background] Wagner SL, White N, Fyfe T, Matthews LR, Randall C, Regehr C, White M, Alden LE, Buys N, Carey MG, Corneil W, Fraess-Phillips A, Krutop E, Fleischmann MH. Systematic review of posttraumatic stress disorder in police officers following routine work-related critical incident exposure. Am J Ind Med. 2020 Jul;63(7):600-615. doi: 10.1002/ajim.23120. Epub 2020 May 17. PMID 32419181
- [Background] Wang WC, Zhang AL, Rasmussen B, Lin LW, Dunning T, Kang SW, Park BJ, Lo SK. The effect of Tai Chi on psychosocial well-being: a systematic review of randomized controlled trials. J Acupunct Meridian Stud. 2009 Sep;2(3):171-81. doi: 10.1016/S2005-2901(09)60052-2. PMID 20633489
- [Background] White-Traut R, Watanabe K, Pournajafi-Nazarloo H, Schwertz D, Bell A, Carter CS. Detection of salivary oxytocin levels in lactating women. Dev Psychobiol. 2009 May;51(4):367-73. doi: 10.1002/dev.20376. PMID 19365797
- [Derived] Dale LP, Dana AN, Lamont H, Nazarloo P, Carter CS, Porges SW, Cuffe SP, Van Vleet Goelz D. Somatic Psychoeducational Intervention Is Associated with Increased Oxytocin Levels, Improved Autonomic Function, and Reduced Psychological Distress Symptoms in Medical and Social Care Professionals. Healthcare (Basel). 2025 Dec 10;13(24):3236. doi: 10.3390/healthcare13243236. PMID 41464305